CLINICAL TRIAL: NCT03881358
Title: Orthokeratology for High Myopia (OHM) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Queensland University of Technology (Other); Aston University (Other)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20180322002
Record Dates: First submitted 2019-02-21; First posted 2019-03-19 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Myopia; High Myopia
Keywords: Myopia control; Orthokeratology; Children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ortho-k lenses and thinner spectacles (Active Comparator): participants using conventionally designed ortho-k lenses (target for 4.00D) and thinner spectacles during day time
  Interventions: Device: ortho-k lenses and thinner spectacles
- newly designed ortho-k lenses (Experimental): participants using newly designed ortho-k lenses for high myopia (target for full correction)
  Interventions: Device: newly designed ortho-k lenses

INTERVENTIONS:
Device: ortho-k lenses and thinner spectacles — Conventinally designed (Emerald) ortho-k lenses (target for -4.00D) and thinner specs during day time
  Arms: ortho-k lenses and thinner spectacles
Device: newly designed ortho-k lenses — Newly designed (Topaz) ortho-k lenses for high myopia (target for full correction)
  Arms: newly designed ortho-k lenses

SUMMARY:
This project aims to investigate/examine high myopic subjects on full correction ortho-k (using Topaz ortho-k lenses for high myopia) compared to subjects undergoing partial reduction ortho-k and their relationship with myopia and myopic progression.

DETAILED DESCRIPTION:
For many years, commercially-available ortho-k lenses aim to reduce low - moderate myopia. Attempts to use these lenses for reduction of high myopia have been shown to give rise to complications such as corneal staining and lens decentration. Thus, practitioners may choose a more conservative way for high myopic children, that is, offering partial reduction ortho-k. Partial reduction ortho-k is target for 4.00-5.00D reduction and the residual refractive errors will be corrected with single vision spectacles to allow good visual acuity in the daytime. Partial reduction ortho-k has been shown to slow axial elongation in high myopic children, however, the main disadvantage is that the children have to wear spectacles in the daytime to correct residual refraction.

Euclid has recently designed a new lens, Euclid's Topaz, for high myopic children. It is currently commercially available to correct myopia for up to 10 D. However, evidence of its effectiveness for visual correction and slowing AL growth is lacking. While numerous studies have shown that orthokeratology is an effective clinical treatment to slow axial eye growth in children, the exact mechanism underlying this reduction in myopia progression associated with orthokeratology remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Myopia: at least 5.00D in one eye or in both eyes
* Astigmatism: ≤1.50D; with-the-rule astigmatism (axes 180 ± 30) ≤1.25D; astigmatism of other axes ≤0.50D in both eyes
* Anisometropia: not be more than 1.00D in the former and not more than 2.00D in the latter.
* Best-corrected Monocular Snellen visual acuity 6/7.5 or better

Exclusion Criteria:

* Strabismus at distance or near
* Previous experience in contact lens wear or myopia control treatment (e.g. refractive therapy or progressive spectacles)
* Contraindication for contact lens wear and orthokeratology (e.g. limbus to limbus corneal cylinder and dislocated corneal apex)
* Previous history of ocular surgery, trauma, or chronic ocular disease
* Concurrent use of medications that may affect tear quality or contact lens wear
* Systemic or ocular conditions that may affect tear quality or contact lens wear (e.g allergy and concurrent medication) or that may affect refractive development (e.g Down syndrome, ptosis)
* Poor compliance to tests (e.g poor fixation in noncontact tonometry or intolerance of lens wear)
* Not willing to comply with the allocated treatment, use and care of lenses and follow-up schedule

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2018-08-04 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in axial length elongation over 24 months. | 2 years
  To determine the change in axial length measured at baseline and two years after lens wear using IOLMaster

SECONDARY OUTCOMES:
First fit success rate of a newly designed ortho-k lens for high myopic children | 1 month
  The success rate in using the first pair of lenses to achieve target refractive correction will be determined
Quality of life (questionnaire) | 3 months
  Quality of life will be determined by questionnaires (using revised Pediatric Refractive Error Profile (PREP) 1 in traditional Chinese version) before and after ortho-k in the two groups of subjects
Ocular aberration | 2 years
  Ocular aberration will be measured by Complete Ophthalmic Analysis System (COAS) aberrometer

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lam CS, Goldschmidt E, Edwards MH. Prevalence of myopia in local and international schools in Hong Kong. Optom Vis Sci. 2004 May;81(5):317-22. doi: 10.1097/01.opx.0000134905.98403.18. PMID 15181356
- [Background] Walline JJ, Lindsley K, Vedula SS, Cotter SA, Mutti DO, Twelker JD. Interventions to slow progression of myopia in children. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD004916. doi: 10.1002/14651858.CD004916.pub3. PMID 22161388
- [Background] Kakita T, Hiraoka T, Oshika T. Influence of overnight orthokeratology on axial elongation in childhood myopia. Invest Ophthalmol Vis Sci. 2011 Apr 6;52(5):2170-4. doi: 10.1167/iovs.10-5485. PMID 21212181
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Swarbrick HA. Orthokeratology review and update. Clin Exp Optom. 2006 May;89(3):124-43. doi: 10.1111/j.1444-0938.2006.00044.x. PMID 16637967
- [Background] Walline JJ, Jones LA, Sinnott LT. Corneal reshaping and myopia progression. Br J Ophthalmol. 2009 Sep;93(9):1181-5. doi: 10.1136/bjo.2008.151365. Epub 2009 May 4. PMID 19416935
- [Background] Charm J, Cho P. High myopia-partial reduction orthokeratology (HM-PRO): study design. Cont Lens Anterior Eye. 2013 Aug;36(4):164-70. doi: 10.1016/j.clae.2013.02.012. Epub 2013 Mar 18. PMID 23518209
- [Background] Cho P, Cheung SW, Edwards MH. Practice of orthokeratology by a group of contact lens practitioners in Hong Kong. Part 2: orthokeratology lenses. Clin Exp Optom. 2003 Jan;86(1):42-6. doi: 10.1111/j.1444-0938.2003.tb03056.x. PMID 12568650
- [Background] Lee TT, Cho P. Relative peripheral refraction in children: twelve-month changes in eyes with different ametropias. Ophthalmic Physiol Opt. 2013 May;33(3):283-93. doi: 10.1111/opo.12057. PMID 23662961
- [Background] Atchison DA, Li SM, Li H, Li SY, Liu LR, Kang MT, Meng B, Sun YY, Zhan SY, Mitchell P, Wang N. Relative Peripheral Hyperopia Does Not Predict Development and Progression of Myopia in Children. Invest Ophthalmol Vis Sci. 2015 Sep 1;56(10):6162-70. doi: 10.1167/iovs.15-17200. PMID 26397463
- [Background] Hiraoka T, Matsumoto Y, Okamoto F, Yamaguchi T, Hirohara Y, Mihashi T, Oshika T. Corneal higher-order aberrations induced by overnight orthokeratology. Am J Ophthalmol. 2005 Mar;139(3):429-36. doi: 10.1016/j.ajo.2004.10.006. PMID 15767050
- [Background] Gonzalez-Meijome JM, Villa-Collar C, Queiros A, Jorge J, Parafita MA. Pilot study on the influence of corneal biomechanical properties over the short term in response to corneal refractive therapy for myopia. Cornea. 2008 May;27(4):421-6. doi: 10.1097/ICO.0b013e318164e49d. PMID 18434845